CLINICAL TRIAL: NCT00841919
Title: Basal/Bolus Insulin Therapy in the Hospital Ward Comparison of Two Protocols: Feasibility Study
Brief Title: Insulin Therapy in the Hospital Comparing Two Protocols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Leon Fogelfeld, John H. Stroger Jr. Hospital of Cook County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBJHS200901
Record Dates: First submitted 2009-02-09; First posted 2009-02-12 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Inpatient; Insulin; Insulin pen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine; Insulin, Isophane; Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): The active control group will receive twice daily NPH insulin as basal insulin and bolus (prandial) insulin as regular insulin to be administered 30 minutes before meals. The administration of basal (prandial) regular insulin and food will be done as the current usual care on the hospital ward. The protocol for initial insulin dose and subsequent dose adjustment has been developed by the "Inpatient Diabetes Advisory Group" and is detailed in appendix B. The patient will receive information regarding diabetes treatments, appropriate diet and diabetic self management which will be provided by the nursing and nutritional staff.
  Interventions: Drug: NPH insulin and regular insulin
- 1 (Experimental): The study group will receive Insulin Glargine as basal insulin and bolus (prandial) insulin as lispro insulin (choice between pens or vials will be made). The administration of bolus (prandial) insulin pen or syringe will be delivered concurrently with the food tray (the concept of "insulin pen/syringe on the food tray") by the nursing staff that together with hospital food services identifies the food tray for the patients in the study group. The protocol for initial insulin dose and subsequent dose adjustment has been developed by the "Inpatient Diabetes Advisory Group" and is detailed in appendix A. The patient will receive information regarding diabetes treatments, appropriate diet and diabetic self management which will be provided by the nursing and nutritional staff
  Interventions: Drug: Glargine insulin; Drug: lispro insulin

INTERVENTIONS:
Drug: Glargine insulin — The study group will receive Insulin Glargine as basal insulin. The protocol for initial insulin dose and subsequent dose adjustment has been developed by the "Inpatient Diabetes Advisory Group" and is detailed in appendix A. The patient will receive information regarding diabetes treatments, appropriate diet and diabetic self management which will be provided by the nursing and nutritional staff.
  Other Names: Lantus insulin
  Arms: 1
Drug: NPH insulin and regular insulin — The active control group will receive twice daily NPH insulin as basal insulin and bolus (prandial) insulin as regular insulin to be administered 30 minutes before meals. The administration of basal (prandial) regular insulin and food will be done as the current usual care on the hospital ward. The protocol for initial insulin dose and subsequent dose adjustment has been developed by the "Inpatient Diabetes Advisory Group" and is detailed in appendix B. The patient will receive information regarding diabetes treatments, appropriate diet and diabetic self management which will be provided by the nursing and nutritional staff.
  Arms: 2
Drug: lispro insulin — Bolus (prandial) insulin as lispro insulin (choice between pens or vials will be made). The administration of bolus (prandial) insulin pen or syringe will be delivered concurrently with the food tray (the concept of "insulin pen/syringe on the food tray") by the nursing staff that together with hospital food services identifies the food tray for the patients in the study group. The protocol for initial insulin dose and subsequent dose adjustment has been developed by the "Inpatient Diabetes Advisory Group" and is detailed in appendix A. The patient will receive information regarding diabetes treatments, appropriate diet and diabetic self management which will be provided by the nursing and nutritional staff.
  Arms: 1

SUMMARY:
The purpose of this study is to determine if by using insulin analog (Glargine and lispro insulin) with an insulin pen the investigators are able to obtain a higher rate of correct timing of insulin and food administration as when compared to the usual therapy (insulin NPH and regular) with syringes.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled blood sugar:

  * Random blood sugar ≥ 200mg/dl
  * Pre-prandial blood sugar greater than 180 mg/dl on two occasions within 24 hours.
* Patient may be off insulin or on subcutaneous inpatient insulin regimen less than 36 hours.
* Transition from an Insulin Drip in the intensive care units to subcutaneous insulin upon transfer to general ward.
* Patient is able to eat and oral feeding is expected.

Exclusion Criteria:

* Patients receiving inpatient oral hypoglycemic agents
* Patients with chronic kidney disease stages 4 & 5 (estimated GFR of <30ml/min) and on dialysis
* Patient with chronic liver disease
* Patient with hypoglycemia unawareness
* Pregnancy
* Patients who are on "NPO" for medical reasons.
* Patient is expected to stay in the hospital for less than 3 days.
* Patient on a new inpatient insulin regimen for > 36 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The rate of correct timing of insulin and food administration | Correct time was 30 min before to 30 minutes after meal was given for control group, and 15 minutes before to 15 minutes after in case group
Pre and post- prandial glucose levels | Pre prandial glucose levels were obtained from 0 to 15 minutes before meal , post prandial glucose levels were obtained 2 hours after mealtime

SECONDARY OUTCOMES:
Length of hospital stay | Measured 24 hours after patient is dischargerd, from day 1 of admission until day of discharge
Nursing staff satisfaction scores for evaluation of the two methods | 24 hours after last patient is discharged
Hypoglycemia rates. | From day 1 of admission until day of discharge, obtained from capillary blood checks done QAC and 2 hours postprandial
High excursions of blood sugars (>300 mg/dl). | From day 1 of admission until day of discharge, obtained from capillary blood checks done QAC and 2 hours postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Leon Fogelfeld, MD, Principal Investigator — John H Stroger Jr. Hospital; Evelyn Lacuesta, MD, Study Chair — John H Stroger Jr. Hospital; Yannis Guerra, MD, Study Chair — Rush University Hospital
Locations (1):
- John H Stroger Jr. Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] Guerra YS, Lacuesta EA, Yrastorza R, Miernik J, Shakya N, Fogelfeld L. Insulin injections in relation to meals in the hospital medicine ward: comparison of 2 protocols. Endocr Pract. 2011 Sep-Oct;17(5):737-46. doi: 10.4158/EP10358.OR. PMID 21454236